CLINICAL TRIAL: NCT00171002
Title: A Multicenter Trial to Evaluate the Safety and Efficacy of the Combination of Valsartan/Amlodipine 160/10 mg Versus Amlodipine 10 mg Alone for 8 Weeks in Hypertensive Patients Who Are Not Adequately Controlled on Amlodipine 10 mg Monotherapy
Brief Title: Efficacy and Safety of Valsartan/Amlodipine Combination in Hypertensive Patients Not Controlled With Amlodipine Alone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVAA489A2306
Record Dates: First submitted 2005-09-10; First posted 2005-09-15 (Estimated); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Hypertension
Keywords: Hypertension, high blood pressure, valsartan, amlodipine
MeSH Terms: conditions — Hypertension | interventions — Amlodipine, Valsartan Drug Combination

INTERVENTIONS:
Drug: valsartan/amlodipine

SUMMARY:
This study will test the effectiveness and safety of a combination treatment in patients whose blood pressure is not controlled with a single medication

ELIGIBILITY:
Inclusion Criteria:

* Patients with uncomplicated, essential hypertension

Exclusion Criteria:

* Severe hypertension
* History of stroke, myocardial infarction, heart failure, chest pain, abnormal heart rhythm
* Liver, kidney, or pancreas disease
* Insulin dependent diabetes
* Allergy to certain medications used to treat high blood pressure

Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 936 (Actual)
Dates: Start 2004-11; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in diastolic blood pressure after 8 weeks

SECONDARY OUTCOMES:
Change from baseline in systolic blood pressure after 8 weeks
Decrease in diastolic blood pressure of at least 10 mmHg or diastolic blood pressure less than 90 mmHg after 8 weeks
Diastolic blood pressure less than 90 mmHg after 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Multiple Locations, Germany
- Novartis Pharmaceuticals, Basel, Switzerland

REFERENCES:
- [Derived] Schunkert H, Glazer RD, Wernsing M, Yen J, Macarie CE, Vintila MM, Romanova J. Efficacy and tolerability of amlodipine/valsartan combination therapy in hypertensive patients not adequately controlled on amlodipine monotherapy. Curr Med Res Opin. 2009 Nov;25(11):2655-62. doi: 10.1185/03007990903251193. PMID 19751115